CLINICAL TRIAL: NCT06530290
Title: Evaluating the Effect of Mirtazapine on Anxiety in Parkinson's Disease Patients; a Randomized Double-blinded Placebo-controlled Clinical Trial
Brief Title: Evaluating the Effect of Mirtazapine on Anxiety in Parkinson's Disease Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leila Dargahi. PharmD PhD (Other)
Responsible Party: Sponsor-Investigator, Leila Dargahi. PharmD PhD, Professor, Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SBMU.PHNS.REC.1400.130
Record Dates: First submitted 2024-04-22; First posted 2024-07-31 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease; Anxiety
Keywords: Parkinson's disease; Anxiety; Mirtazapine
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirtazapine (Experimental): Mirtazapine (15 mg), once a day, for 12 weeks
  Interventions: Drug: Mirtazapine 15 MG
- Placebo (Placebo Comparator): Placebo, once a day, for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine 15 MG — Mirtazapine (15 mg), once a day for 12 weeks
  Arms: Mirtazapine
Drug: Placebo — Placebo, once a day, for 12 weeks
  Arms: Placebo

SUMMARY:
This study is a single-center, parallel and double-blind study in Movement Disorders Clinic of Shohadaye Tajrish Hospital. Patients, researchers (physicians, outcome assessors) and data analysts are blinded. After assessing the inclusion and exclusion criteria's, patients who assigned the informed consent form, are randomly divided into control and treatment groups.Patients in treatment or placebo groups respectively receive mirtazapine (15 mg) or placebo, once a day for 12 weeks. Primary (anxiety) and secondary (depression, fatigue, sleep disorders, and quality of life) outcomes are evaluated at baseline, and after 4 and 12 weeks of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 17 years old
* Patient with Parkinson's disease according to UKPDSBB criteria
* Patient with mild/moderate Parkinson's disease according to Hoehn and Yahr Scale (HY score = 1-3)
* Self-report or clinical diagnosis of anxiety
* Patients who have signed informed consent to participate in the study.

Exclusion Criteria:

* Pregnant and lactating women
* Parkinson's patients with onset of disease in less than 1 year
* Unstable medication for Parkinson's disease during the last two weeks
* Parkinson's patients with DBS
* Patients with other neurodegenerative diseases like multiple system atrophy (MSA), Huntington's and etc.
* Patients with major depressive disorder
* A history of using SSRIs, SNRIs, benzodiazepines and β-blockers during the last 4 weeks
* A history of using MAO inhibitors
* A history of alcohol and substance abuse
* A history of acute stress during the last 3 months
* A history of suicide
* A history of cardiovascular diseases
* A history of liver and or kidney disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety score | Baseline, and after 4 and 12 weeks of treatment
  Anxiety score using Hamilton Anxiety Rating Scale (HAM-A)
Anxiety score | Baseline, and after 4 and 12 weeks of treatment
  Parkinson Anxiety Scale (PAS) questionnaires

SECONDARY OUTCOMES:
Depression score | Baseline, and after 4 and 12 weeks of treatment
  Depression score using Hamilton Depression Rating Scale (HAM-D) questionnaire
Fatigue score | Baseline, and after 4 and 12 weeks of treatment
  Fatigue score using Parkinson's Disease Fatigue Scale (PDFS) questionnaire
Sleep disorder score | Baseline, and after 4 and 12 weeks of treatment
  Sleep disorder score using Parkinson's disease Sleep Scale (PDSS) questionnaire
Quality of life score | Baseline, and after 4 and 12 weeks of treatment
  Quality of life score using Parkinson's Disease Quality of Life (PDQL) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Leila Dargahi, PharmD/PhD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Mehri Salari, MDFellowship, Principal Investigator — Shahid Beheshti University of Medical Sciences; Neda Valian, PhD, Study Director — Shahid Beheshti University of Medical Sciences; Leila Mohaghegh Shalmani, PharmD/PhD, Study Chair — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid Beheshti University of Medical Sciences, Shohada-e-Tajrish Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No